CLINICAL TRIAL: NCT00664105
Title: PhII Study of Concurrent Chemoradiotherapy With Weekly Docetaxel, Carboplatin and Radiation Therapy Followed by Consolidation Chemotherapy With Docetaxel and Carboplatin for Locally Advanced Inoperable Non-small Cell Lung Cancer (NSCLC)
Brief Title: Ph II Concurrent Chemo t/Docetaxel/Carboplatin/Radio Therapy-consolidation t/Locally Adv Inoperable Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment became standard.
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vicki Keedy, MD, Assistant Professor of Medicine; Clinical Director, Sarcoma Program; Assistant Medical Director, Clinical Trials Shared Resource; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 0319; VU-VICC-THO-0319; VU-VICC-030269
Record Dates: First submitted 2008-04-19; First posted 2008-04-22 (Estimated); Results first posted 2011-03-22 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be given weekly for seven weeks beginning on Day 1 of the study as a 30-minute intravenous infusion during concurrent therapy.
  Carboplatin will be given once every three weeks as a 30-minute intravenous infusion immediately following the infusion of docetaxel. Patients will receive two cycles of consolidation treatment.
  Other Names: None specified
Drug: Docetaxel — Docetaxel will be given weekly for seven weeks beginning on Day 1 of the study as a 30-minute intravenous infusion during concurrent therapy.
  Docetaxel will be given once every three weeks administered as a one-hour IV infusion. Patients will receive two cycles of consolidation treatment (1 cycle = 3 weeks).
  Other Names: Taxotere
Radiation: radiation therapy — Radiotherapy will be administered daily X 5 day/week for 34 days beginning on Day 1 of the study. Radiotherapy will follow immediately after the infusions of docetaxel and carboplatin.
  Other Names: none specified

SUMMARY:
RATIONALE: Because of its success in advanced NSCLC both as a single agent and in combination with other chemotherapeutics, it is reasonable to investigate the efficacy and toxicity of docetaxel as a multimodality regimen in this patient population. Docetaxel at a dose of 20 mg/m2 appears to be a well-tolerated "weekly" dose when combined with either cisplatin 25 mg/m2 20-22 or carboplatin area under the curve (AUC) 2 23-25 concomitant with radiation therapy.

PURPOSE: To explore the potential benefits of the radiosensitizing effects of weekly docetaxel/carboplatin/radio therapy concurrent therapy followed full dose systemic docetaxel/carboplatin consolidation therapy on overall response rate, survival, progression-free survival, safety and toxicity in patients with locally advanced NSCLC.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall survival (0S) for advanced NSCLC patients receiving concurrent chemoradiotherapy with weekly docetaxel, carboplatin and radiation therapy followed by two cycles of consolidation chemotherapy with docetaxel and carboplatin.

Secondary

* To determine the overall response rate in patients treated with this regimen.
* To determine the time to disease progression in patients treated with this regimen.
* To assess the safety and tolerability of this regimen in these patients.

OUTLINE:

* This is a Phase II, open label, multi-center study to determine the overall survival rate for patients treated with concurrent chemoradiotherapy with weekly docetaxel, carboplatin and radiation followed by two cycles of consolidation chemotherapy with docetaxel and carboplatin. Eligible patients will receive concurrent therapy with docetaxel (20 mg/m2) administered weekly for seven weeks as a 30-minute intra-venous (IV) infusion followed by carboplatin (AUC 2) administered weekly for seven weeks as a 30-minute IV infusion. Concurrent radiation therapy will be administered at a dose of 1.8 Gy daily 5 days/week for 25 fractions followed by a dose of 2.0 Gy daily, 5 days/week for 9 fractions (total of 34 fractions). There will be a three-week rest period following the end of the concurrent chemotherapy after which the consolidation phase will begin. During this phase of the study, patients will be treated with docetaxel (75 mg/m2) administered as a 1-hour IV infusion followed by carboplatin (AUC 6) administered as a 30-minute IV infusion. Patient will be treated every three weeks for a total of two cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must voluntarily sign and date an informed consent before the initiation of any study procedures
* Patients must have non-metastatic, inoperable, Stage IIIA or IIIB histologically or cytologically documented NSCLC without evidence of malignant pleural effusion
* Patients must not have received any prior systemic chemotherapy, thoracic radiotherapy or surgical resection for treatment of NSCLC
* Patients must have at least one site of unidirectionally measurable disease
* Patients must be ≥ 3 weeks from a formal exploratory thoracotomy
* Patients must have a Radiation Oncology and Medical Oncology consult and approval prior to study entry
* Patients must be ≥ 18 years of age
* Women of childbearing potential must have a negative baseline serum pregnancy within 7 days prior to Week 1, Day 1 and must not be breast feeding.
* Women of childbearing potential and men with a sexual partner of child bearing potential must use an effective method of contraception beginning prior to study entry, for the duration of the study participation and for a minimum of 3 months after the last dose of chemotherapy.
* Patients must have adequate hepatic, renal, lung and bone marrow function as defined below:

  * Absolute neutrophil count (ANC) > 1,500/mm3
  * Hemoglobin > 9.0 gm/dL
  * Creatinine < 1.5
  * Platelets > 100,000/mm3
  * Total bilirubin within normal limits (WNL)
  * AST or ALT and Alkaline Phosphatase must be within the range allowing for eligibility, as per chart on page 10 of the protocol.
* Calculated CrCl > 50 ml/min (via Cockroft-Gault formula).
* Forced expiratory volume in 1 second (FEV 1) > 800 ml

Exclusion Criteria:

* Known hypersensitivity to drugs formulated with polysorbate 80
* Peripheral neuropathy Grade ≥ 2.
* Wet stage IIIB (documented malignant pleural effusion) or stage IV NSCLC
* Previous chemotherapy or radiation therapy
* Any concomitant malignancy, brain metastasis or uncontrolled, clinically significant medical or psychiatric disorder
* Pregnant or nursing women
* A greater than or equal to 10% weight loss over the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Keedy, MD, Study Director — Vanderbilt-Ingram Cancer Center
Locations (15):
- United States (15):
  - M.D. Anderson Cancer Center, Orlando, Orlando, Florida
  - Chesapeake Oncology Hematology Associates, Baltimore, Maryland
  - University Hospital of Cleveland, Cleveland, Ohio
  - Lehigh Valley Hospital - John & Dorothy Morgan Cancer Center, Allentown, Pennsylvania
  - Erlanger Health System, Chattanooga, Tennessee
  - Clarksville Regional Hematology Oncology Group, Clarksville, Tennessee
  - Jackson Madison County Hospital, Jackson, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - The West Clinic, PC, Memphis, Tennessee
  - St. Thomas Health Services, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period = 2/18/2004 through 1/23/2007
Pre-assignment Details: A total of 66 people consented to take part in this study and of those, 1 was determined to be ineligible and 2 withdrew from the study prior to beginning protocol therapy.
Groups:
- Chemo-radio Therapy: Patients will receive carboplatin and docetaxel will be given weekly for seven weeks during concurrent radiotherapy. After a 3-week rest, patients will receive treatment every 3 weeks for two cycles of consolidation treatment.
Period: Overall Study
Arm/Group | Chemo-radio Therapy
Started | 63
Completed | 39
Not Completed | 24
Not completed — Death | 3
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 9
Not completed — Disease progression | 7

BASELINE CHARACTERISTICS:
Arm/Group | Chemo-radio Therapy
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Months from on-study to expired/last date known alive.
Time Frame: 14.95 months (average duration, on study date to off-study date)
Population: Patients who received at least one treatment and who were available for determination of overall survival.
Measure: Median (Full Range); unit: Months
Arm/Group | Chemo-radio Therapy
Number analyzed (Participants) | 63
Months | 11 [0 to 47]

2. Secondary Outcome: Overall Response Rate
Description: Patient response to treatment per RECIST:
  Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started Complete response (CR): disappearance of all target lesions Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD
Time Frame: on-study date to date of best response
Population: Patients who were available for measurement of response. Six patients were not available for measurement of response and are not included in the analyzed population
Measure: Number; unit: participants
Groups:
- Chemo-radio Therapy: Patients will receive carboplatin and docetaxel weekly for seven weeks during concurrent radiotherapy. After a 3-week rest, patients will receive treatment every 3 weeks for two cycles of consolidation treatment.
Arm/Group | Chemo-radio Therapy
Number analyzed (Participants) | 57
participants
  Complete Response | 6
  Partial Response | 33
  Progressive Disease | 5
  Stable Disease | 13

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression in months
Time Frame: on-study date to date of progression
Population: Patients with disease progression.
Measure: Median (Full Range); unit: Months
Arm/Group | Chemo-radio Therapy
Number analyzed (Participants) | 39
Months | 5 [1 to 25]

4. Secondary Outcome: Number of Participants With Adverse Events by Grade
Description: Number of participants with adverse events, according to grade of event, using the NCI Common Toxicity Criteria (version 2.0) grading system to assign a grade to each event with 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, and 5 = death related to adverse event
Time Frame: 30 days after last treatment.
Population: Patients who received treatment and who experienced an adverse event.
Measure: Number; unit: participants
Arm/Group | Chemo-radio Therapy
Number analyzed (Participants) | 63
participants
  Grade 1 | 11
  Grade 2 | 19
  Grade 3 | 35
  Grade 4 | 12
  Grade 5 | 3

ADVERSE EVENTS:
Arm/Group | Chemo-radio Therapy
Serious Adverse Events (participants affected / at risk) | 37/63
Other Adverse Events (participants affected / at risk) | 13/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo-radio Therapy (N=63)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Bleeding (associated with surgery) (Surgical and medical procedures) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Infection Other, Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 8 (10)
Depressed level of consciouness (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysphagia - pharynegal (related to radiation) (Gastrointestinal disorders) | 1 (1)
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 14 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fainting (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hemoglobin decrease (Investigations) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3)
Mucositis (due to radiation) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Neutrophil count decrease (Investigations) | 2 (2)
Pain due to radiation (Surgical and medical procedures) | 1 (1)
Infection other, peg tube abcess (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Supraventricular arrhythmias (Cardiac disorders) | 2 (2)
Transfusion: Packed-Red-Blood-Cells (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Investigations) | 6 (6)
Incomplete fracture of right humerus (Musculoskeletal and connective tissue disorders) | 1 (1)
pericardial effusion (Cardiac disorders) | 1 (1)
Thrombosis (Cardiac disorders) | 6 (7)
Hemorrhage, upper GI bleed (Gastrointestinal disorders) | 1 (1)
Infection without neutropenia (Metabolism and nutrition disorders) | 5 (5)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo-radio Therapy (N=63)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
Fever (General disorders) | 3 (4)
Dehydration (Musculoskeletal and connective tissue disorders) | 3 (3)
Weight loss (Investigations) | 5 (5)

LIMITATIONS AND CAVEATS:
Outcome measure #4, "Number of participants with AEs by grade", will not match the total number of participants in this study. Some participants have multiple events in one or more grade designations or some participants have no events at all.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes